CLINICAL TRIAL: NCT04758221
Title: Clinical Performance of Composite Coronal Build -Up in Mutilated Primary Incisors: Prospective Single Arm Study
Brief Title: Clinical Performance of Composite Coronal Build -Up in Mutilated Primary Incisors: 3 Years Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Associate Professor Dr. Rania Abdallah Nasr, Associate Professor Dr. Rania Nasr, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41720
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Early Childhood Caries; Pediatric Disease; Dental Caries; Dental Diseases
Keywords: Child; Esthetics; Dental caries; Primary incisors; Composite
MeSH Terms: conditions — Dental Caries; Stomatognathic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm : Composite coronal build up strip crown (Experimental): A total of (42) decayed or traumatized primary anterior teeth were treated with composite coronal build-up based on the micromechanical adhesive procedure of composite resin in addition to macro mechanical retentive grooves created on the lateral sides of the cervical one third of the roots of treated teeth.
  Interventions: Other: Treatment by composite coronal build-up

INTERVENTIONS:
Other: Treatment by composite coronal build-up — A total of (42) decayed or traumatized primary anterior teeth were treated with composite coronal build-up based on the micromechanical adhesive procedure of composite resin in addition to macro mechanical retentive grooves created on the lateral sides of the cervical one third of the roots of treated teeth.

SUMMARY:
Prospective single arm study was to evaluate the clinical success and/ or failure of resin-bonded composite coronal build-up retained by macro-retentive grooves for restoring mutilated primary maxillary incisors after 36 months.

Design: Forty two primary incisors out of 14 children, aged 2-5years, treated in a private pediatric dental practice under general anesthesia and presented for follow-up after 6, 12, 18, 24 and 36 months included in the study. The parameters recorded at the baseline and at the follow-up intervals were: retention, colour match, the number and location of the decayed surfaces (recurrent caries), chipping /fracture of the restoration and loss of restoration (failure).

Materials and Methods: A total of (14) pediatric patients aged from 2-5 years presented with mutilated primary anterior teeth due to caries or trauma and treated comprehensively under general anesthesia from June 2016 to June 2017 were enrolled in this study. A total of (42) decayed or traumatized primary anterior teeth were treated with composite coronal build-up based on the micro-mechanical adhesive procedure of composite resin in addition to macro mechanical retentive grooves created on the lateral sides of the cervical one third of the roots of treated teeth. The patients returned at the end of 6, 12, 18, 24 and 36 months and received clinical examinations. Another dentist (co-author) who did not attend the treatment evaluated the strip crowns clinically by modified United States Public Health Service (USPHS) criteria.

DETAILED DESCRIPTION:
Purpose: The purpose of this study was to evaluate the clinical success and/ or failure of resin-bonded composite coronal build-up retained by macro-retentive grooves for restoring mutilated primary maxillary incisors after 36 months.

Design: Forty two primary incisors out of 14 children, aged 2-5years, treated in a private pediatric dental practice under general anesthesia and presented for follow-up after 6, 12, 18, 24 and 36 months included in the study. The parameters recorded at the baseline and at the follow-up intervals were: retention, colour match, the number and location of the decayed surfaces (recurrent caries), chipping /fracture of the restoration and loss of restoration (failure).

Materials and Methods: A total of (14) pediatric patients aged from 2-5 years presented with mutilated primary anterior teeth due to caries or trauma and treated comprehensively under general anesthesia from June 2016 to June 2017 were enrolled in this study. A total of (42) decayed or traumatized primary anterior teeth were treated with composite coronal build-up based on the micromechanical adhesive procedure of composite resin in addition to macro mechanical retentive grooves created on the lateral sides of the cervical one third of the roots of treated teeth. The patients returned at the end of 6, 12, 18, 24 and 36 months and received clinical examinations. Another dentist (co-author) who did not attend the treatment evaluated the strip crowns clinically by modified United States Public Health Service (USPHS) criteria. The USPHS system is primarily for posterior teeth, so a new system was developed for anterior teeth. The definitions and criteria for the rating system are detailed in Table (1). Briefly, it was a photographic examination including an evaluation of the color, shape, and integrity of the strip crown.

All patients were recalled, and restorations were evaluated for anatomic form, surface texture, recurrent caries, color match and retention in accordance with Ryge's Direct (US Public Health Service) evaluation criteria at baseline (immediately postoperative), and intervals of 6, 12, 24, and 36 months.

The crown was considered to be clinically successful, if the surface appeared smooth, the colour remained good or acceptable, without chipping/ fracture or recurrent caries at tooth/restoration interface and there is no loss of the restoration.

Data are analyzed using percentages, frequencies and cumulative frequencies. The Z-test will be used for comparison between failure rates of the two types of failures (Failure due to trauma & failure of bonding), significance level is set at P< 0·05. The Chi squared test will be used for association between the number of affected surfaces and the total failures. The level of significance (P-value) is set at P< 0·05.

ELIGIBILITY:
Inclusion Criteria:

* Only children in the age group of 2-5 years.

  * Teeth affected due to caries or trauma with one or two or three surfaces affected or more.

Exclusion Criteria:

* • Any tooth nearing exfoliation or not fit for restoration.

  * Patients with systemic problems which may interfere with general anesthesia.
  * Teeth with excessive pathologic mobility.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical performance of composite strip crowns. | 36 months
  Evaluation of the clinical performance of composite strip crowns. By Clinical photographs.

SECONDARY OUTCOMES:
Assessment of success and failure of the composite coronal build-up after 3 years follow-up. | 36 months
  Assessment of success and failure of the composite coronal build-up after 3 years follow-up in terms of:
  * Retention
  * Color match
  * Recurrent Caries
  * Fracture/Chipping
  * Loss of restoration (Failure)

CONTACTS AND LOCATIONS:
Overall Officials: Rania Nasr, Assoc. Prof., Principal Investigator — Faculty of Dentistry, Cairo University, Egypt
Locations (1):
- Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
No sharing of any private data of participants with other researchers